CLINICAL TRIAL: NCT05058976
Title: Innovative Approach to Geriatric Osteoporosis
Brief Title: Romosozumab Use to Build Skeletal Integrity
Acronym: RUBI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Susan L. Greenspan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Susan L. Greenspan, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20060028; 5R01AG066825-02 (NIH)
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal; Osteoporosis Fracture
Keywords: Bone loss; Nursing Home Patients; Long-term Care Patients; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Osteoporotic Fractures; Bone Diseases, Metabolic | interventions — romosozumab; Zoledronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Romosozumab, then Zoledronic Acid (Experimental): Monthly dose: 210 mg Romosozumab subcutaneous injections; Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplements); all participants will receive 5 mg Zoledronic Acid IV infusion at the Month 12 visit.
  Interventions: Drug: Romosozumab; Drug: Zoledronic acid; Dietary Supplement: Calcium and Vitamin D
- Placebo, then Zoledronic Acid (Placebo Comparator): Monthly dose: placebo saline subcutaneous injections; Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplements); all participants will receive 5 mg Zoledronic Acid IV infusion at the Month 12 visit.
  Interventions: Drug: Placebo; Drug: Zoledronic acid; Dietary Supplement: Calcium and Vitamin D

INTERVENTIONS:
Drug: Romosozumab — Monthly dose: 210 mg subcutaneous injection
  Other Names: Evenity
  Arms: Romosozumab, then Zoledronic Acid
Drug: Placebo — Monthly saline injection
  Arms: Placebo, then Zoledronic Acid
Drug: Zoledronic acid — 5 mg IV infusion at Month 12 Visit
  Other Names: Reclast
Dietary Supplement: Calcium and Vitamin D — Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplement)

SUMMARY:
The purpose of this study is to find out if one year of romosozumab (Evenity®), a monthly injection given in the arm under the skin, prior to an infusion of zoledronic acid Reclast®, works to treat bone loss and prevent it from worsening in older women (ages 65 and older) who have osteoporosis and reside in long-term care (LTC) facilities.

DETAILED DESCRIPTION:
Objective:

The long-term goal of this study is to improve health, well-being and quality of life in the frail Long-term Care (LTC) population by reducing fractures. The short-term goal is to demonstrate efficacy of the novel dual action Romosozumab (ROMO) to improve Bone Mineral Density (BMD) and skeletal integrity and its safety, a necessary (but not sufficient) precondition of a large fracture reduction trial. The investigators propose to conduct a 2-year, randomized, double-blind, calcium vitamin D controlled trial to test the efficacy and safety of the sclerostin inhibitor ROMO among a cohort of 200 underserved, institutionalized, frail women ≥65 years old. Bone measures will be collected in a mobile lab. The monthly subcutaneous therapy negates concerns regarding poor oral absorption or compliance. The use of annual Zoledronic Acid (ZOL) to follow ROMO, will prevent bone loss and insure the entire group will be provided with at least 1 year of therapy. The groups include: 1) ROMO →ZOL vs 2) placebo →ZOL.

Aim 1: Evaluate efficacy of bone building ROMO treatment prior to ZOL in improving bone mineral density. H1: Women on ROMO →ZOL will have greater hip and spine BMD increases after 2 years (H1.1-primary) and 1 year (H1.2), and at other locations (H1.3).

Aim 2: Examine improvements in 3D trabecular microstructure (TBS), markers of bone turnover and collect preliminary evidence for a fracture reduction trial. The investigators will measure vertebral trabecular bone score (TBS), a 3-D microarchitectural image and parameters of the spine, hip, and lateral spine H2: Women on ROMO →ZOL will have greater increases in TBS measures of spine, hip and lateral spine after one (H2.1) and two (H2.2) years; and improvement in bone turnover markers (CTx and P1NP; H2.3).

Aim 3: Determine characteristics associated with responders and non responders. The investigators will use multiple regression analyses and other data mining techniques to identify baseline characteristics of responders and non-responders. H3.1: Poor baseline functional/cognitive status/immobility will be associated with poor bone healthy outcomes. H3.2: Greater early changes in bone turnover markers will be associated with greater skeletal improvements.

ELIGIBILITY:
Inclusion Criteria:

Elderly women 65 years and older will be considered if:

* They reside in an institution (nursing home or assisted living facility or senior care community);
* They have a) osteoporosis by axial bone density (spine, hip or forearm BMD T-score≤ -2.5 SD), b) a previous adult fragility fracture of the spine or hip or c) would be treated based on FRAX and the National Osteoporosis Foundation (NOF) treatment thresholds of a 10 year risk of 10% for a major osteoporotic fracture or ≥ 3% for hip fracture using femoral neck BMD.
* Willing and able to complete the informed consent process or provide consent by proxy.

Exclusion Criteria:

* Those with subacute illnesses who are not expected to survive or who will be discharged in less than 2 years.
* Those who have previously had an acute cardiovascular or cerebrovascular event within the preceding year. specifically, no recent history of coronary heart disease, heart failure, significant arrhythmia, stroke or Transient Ischemic Attack (TIA).
* Recent cardiovascular disease (CVD) symptoms (significant chest pain, congestive heart failure, shortness of breath, or palpitations or cerebrovascular symptoms such as numbness or weakness in the face, arm, legs, difficulty talking, changes in vision, loss of balance, headache, feeling light-headed or dizzy).
* Unstable angina.
* Those who are currently on therapy (including a bisphosphonate, denosumab, teriparatide, abaloparatide or romosozumab) or have been on a bisphosphonate for greater than 1 year during the previous 2 years.
* Those who are unable to take an intravenous bisphosphonate (zoledronic acid) due to renal insufficiency with eGFR < 35 ml/min.
* Vitamin D levels <25 ng/mL.
* Participants will be allowed to continue on medications known to affect bone and mineral metabolism (e.g., glucocorticoids, anticonvulsants) because their use is common in this population.
* Those who have been treated in the past or present with osteoporosis agents, such as estrogen/progesterone or raloxifene will be allowed to participate and continue on these therapies if prescribed by their physician.
* Patients will be allowed to wear hip pads if prescribed by their physician.
* Non-ambulatory residents (those who cannot stand and pivot with assistance in order to transfer to the DXA table) will be excluded.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density of the total hip | 24 months
  Bone Mineral Density (BMD) of the total hip at 24 months as assessed by dual-energy x-ray absorptiometry (DXA)
Bone Mineral Density of the spine | 24 months
  Bone Mineral Density (BMD) of the spine at 24 months as assessed by dual-energy x-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Senior Communities, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared will include all IPD collected, with the exception of essential identifying information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Any data request will be considered only after main planned manuscripts have been accepted for publication.
Access Criteria: The PI and the investigative team will review data requests. If approved, all essential identifying information will be removed prior to data distribution. When a request of the data is received, a data sharing agreement will be sent to the requestor which will specifically include requirements for privacy and confidentiality, especially that no attempt will be made to identify study participants, that the data will not be redistributed, and will be destroyed after completing the specific stated purpose. Upon receipt of the signed data sharing agreement, the PI will send the distribution file to the requestor using an appropriate modality such as email or cloud storage.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT05058976/ICF_000.pdf